CLINICAL TRIAL: NCT05199194
Title: Randomization to EndoVascular Treatment Alone or Preceded by Systemic Thrombolysis With Tenecteplase in Acute Ischemic Stroke Due to Large Intracranial VEssel OcclusioN Trial - DIRECT Thrombectomy vs. Intravenous TNK Plus Thrombectomy
Brief Title: Randomization to Endovascular Treatment Alone or Preceded by Systemic Thrombolysis With Tenecteplase in Ischemic Stroke
Acronym: DIRECT-TNK
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Hospital Moinhos de Vento (Other)
Collaborators: Ministry of Health, Brazil (Other Government); Boehringer Ingelheim (Industry); Medtronic (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RESILIENT DIRECT-TNK
Record Dates: First submitted 2022-01-06; First posted 2022-01-20 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Stroke, Ischemic; Stroke, Acute
Keywords: Tenecteplase; TNK; MT; Mechanical Thrombectomy
MeSH Terms: conditions — Ischemic Stroke; Stroke | interventions — Tenecteplase

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mechanical Thrombectomy preceded by TNK (Experimental): Subjects assigned to this arm will receive an intravenous bolus of tenecteplase (0.25mg/kg) before the mechanical thrombectomy.
  Interventions: Drug: Tenecteplase
- Mechanical Thrombectomy preceded by Placebo (Placebo Comparator): Subjects assigned to this arm will receive an intravenous bolus of matching placebo (with the same volume of infusion as of 0.25mg/kg of tenecteplase) before the mechanical thrombectomy.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tenecteplase — Intravenous thrombolysis with tenecteplase 0.25mg/kg
  Other Names: TNK
  Arms: Mechanical Thrombectomy preceded by TNK
Drug: Placebo — Intravenous administration of placebo, matching the volume of tenecteplase 0.25mg/kg
  Arms: Mechanical Thrombectomy preceded by Placebo

SUMMARY:
A phase III randomized, multi-center, double-blinded, placebo-controlled clinical trial that will examine two strategies for the treatment of acute ischemic stroke associated with a large vessel anterior occlusion within 4.5 hours from symptoms onset: direct endovascular treatment vs. endovascular treatment preceded by intravenous tenecteplase.

DETAILED DESCRIPTION:
Randomized, prospective, multicenter, double-blinded, placebo-controlled clinical trial with adaptive desing. Randomization will be 1:1 according to reperfusion treatment modalities: (A) (with placebo TNK) direct mechanical thrombectomy vs. (B) Intravenous thrombolysis with TNK (0.25 mg/kg) plus mechanical thrombectomy. Randomization will be done by a minimization process using age, National Institute of Health Stroke Scale (NIHSS) score, and site of the occluded artery. For the primary outcome, the subjects will be followed up within 90 days after randomization. The primary outcome will be the ordinal distribution from the modified Rankin scale score (mRS).

Subjects presenting acute ischemic stroke within 4.5 hours of the onset of symptoms attributable to an occlusion of intracranial internal carotid or of the proximal middle cerebral artery (MCA, M1- or M2-segment) with or without tandem occlusion of cervical internal carotid confirmed by vascular neuroimaging. Subjects should be eligible for IV thrombolysis. In the sample size calculation, a difference in treatment effect between the groups (achievement of mRS 0 to 2 at 90 days) of 10.6% was considered, with 33.8% in the intervention group (TNK + thrombectomy) and 23.2% in the control group (placebo + thrombectomy), using a unilateral alpha of 0.025, with a power of 80%, resulting in a sample size of 358 participants. Considering a loss ratio of 10%, a sample size of 398 participants is estimated (199 in each treatment arm). An interim analysis is planned to be executed with 50% and 75% of the total sample. It allows the trial to be terminated in the case of efficacy or futility, in addition to enabling adaptive designed based on conditional probability of a positive result.

ELIGIBILITY:
Inclusion Criteria:

* Acute ischemic stroke where a patient is eligible for IV thrombolytic treatment within 4.5 hours of stroke onset.
* No significant pre-stroke functional disability (mRS ≤ 1)
* Baseline NIHSS scores obtained before randomization must be equal to or higher than 6 points
* Age equal ≥ 18 and =< 85 years
* Occlusion (TICI 0-1) of the ICA or proximal MCA segments (M1 or M2) suitable for endovascular treatment, as evidenced by CTA, MRA, or angiogram, with or without concomitant cervical carotid stenosis or occlusion.
* Patient randomized within 4.5 hours of symptom onset. Symptoms onset is defined as the point in time the patient was last seen well (at baseline). Treatment start is defined as groin puncture, max 90 minutes after randomization.

  * Patients who have woken up with the symptoms and who have a mismatch FLAIR-DWI according to the WAKE-UP Trial will be considered as having a time window of <4.5h.
* Informed consent obtained from the patient or acceptable patient surrogate.

Exclusion Criteria:

* Known hemorrhagic diathesis, coagulation factor deficiency, or oral anticoagulant therapy with INR > 1.7 or direct oral anticoagulants such as thrombin antagonists (ex: dabigatran) or X factor (ex: rivaroxaban, apixaban, edoxaban) at the least 48 hours.
* Baseline platelet count < 100.000/μL
* Baseline blood glucose of < 50mg/dL or > 400mg/dl
* Severe, sustained hypertension (SBP > 185 mm Hg or DBP > 110 mm Hg) NOTE: If the blood pressure can be successfully reduced and maintained at the acceptable level using AHA guidelines recommended medication (including iv antihypertensive drips), the patient can be enrolled.
* Patients in coma (NIHSS item of consciousness >1) (Intubated patients for transfer could be randomized only in case an NIHSS is obtained by a neurologist prior transportation).
* Seizures at stroke onset which would preclude obtaining a baseline NIHSS
* Serious, advanced, or terminal illness with anticipated life expectancy of less than one year.
* History of life-threatening allergy (more than rash) to contrast medium.
* Subjects who has received IV t-PA treatment before the randomization.
* Renal failure with serum creatinine ≥ 3 mg/dl
* Woman of childbearing potential who is known to be pregnant or who has a positive pregnancy test on admission.
* Subject participating in a study involving an investigational drug or device that would impact this study.
* Cerebral vasculitis, endocarditis or subarachnoid hemorrhage.
* Patients with a pre-existing neurological or psychiatric disease that would confound the neurological or functional evaluations.
* Unlikely to be available for 90-day follow-up (e.g. no fixed home address, visitor from overseas).
* Hypodensity on CT more than one third of MCA territory or hypersignal in more than one third of MCA territory on MR-DWI.
* ASPECTS score < 6 (no contrast at least 5 mm cut imaging on CT) or on MR-DWI sequence.
* CT or MR evidence of hemorrhage (the presence of < 5 GRE, SWI, SWAN microbleeds is allowed).
* Significant mass effect with midline shift.
* Evidence of ipsilateral carotid occlusion, high grade stenosis or arterial dissection in the extracranial or petrous segment of the internal carotid artery that cannot be treated or will prevent access to the intracranial clot or excessive tortuosity of cervical vessels precluding device delivery/deployment.
* Subjects with occlusions in multiple vascular territories (e.g., bilateral anterior circulation, or anterior/posterior circulation).
* Evidence of intracranial tumor (except small meningioma).

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 398 (Estimated)
Dates: Start 2022-05-27 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Distribution of the modified Rankin Scale scores at 90 days | 90 days
  Distribution of the modified Rankin Scale scores (shift analysis).

SECONDARY OUTCOMES:
Functional independence defined as modified Rankin Score ≤ 2 | 90 days
  Functional independence defined as modified Rankin Score ≤ 2
Infarct volume evaluated on CT at 24 hours (-2/+12 hours). | 24 hours
  Infarct volume evaluated on CT at 24 hours (-2/+12 hours).
Dramatic early favorable response as determined by a National Institute of Health Stroke Scale (NIHSS) of 0-2 or NIHSS improvement ≥ 10 points at 24 (-2/+12 hours) hours. | 24 hours
  Dramatic early favorable response as determined by a National Institute of Health Stroke Scale of 0-2 or NIHSS improvement ≥ 10 points at 24 (-2/+12 hours) hours.
Cost-effectiveness analysis of endovascular therapy alone vs. endovascular therapy associated with tenecteplase | 12 months
  Cost-effectiveness analysis of endovascular therapy alone vs. endovascular therapy associated with tenecteplase
Quality of life analysis as measured by EuroQol/EQ5D at 3 month, 6 months and one year among the groups | 3 months, 6 months and 12 months
  Quality of life analysis as measured by EuroQol/EQ5D at 3 month, 6 months and one year among the groups
Score distribution of mRS at 90 days (shift analysis) in patients presenting M2-CMA occlusion | 90 days
  Score distribution of mRS at 90 days (shift analysis) in patients presenting M2-CMA occlusion
Vessel recanalization evaluated by CT angiography or MRA at 24 hours in both treatment groups | 24 hours
  Vessel recanalization evaluated by CT angiography or MRA at 24 hours in both treatment groups
Vessel recanalization post procedure in the endovascular arm assessed by TIMI grades and adjudicated by a central core-lab. Successful recanalization is defined as TICI (Thrombolysis in Cerebral Infarction) 2b or 3 on the post-procedure angiogram. | Immediately Post-procedure
  Vessel recanalization post procedure in the endovascular arm assessed by TIMI grades and adjudicated by a central core-lab. Successful recanalization is defined as TICI (Thrombolysis in Cerebral Infarction) 2b or 3 on the post-procedure angiogram.

OTHER OUTCOMES:
Mortality at 90 days | 90 days
  Mortality at 90 days
Mortality related to stroke and complications at 90 days | 90 days
  Mortality related to stroke and complications at 90 days
Clinically significant ICH rates at 24 (-2/+12) hours. | 24 hours
  All intracerebral hemorrhages will be classified by a central core-lab using the ECASS criteria. Symptomatic ICH will be defined as per the SITS-MOST definition: deterioration in NIHSS score of ≥4 points within 24 hours from treatment and evidence of intraparenchymal hemorrhage type 2 in the 22 to 36 hours follow-up imaging scans. The incidence of any asymptomatic hemorrhage measured at 24 (-2/+12) hours will also be compared.
Procedural related complications | 7 days
  arterial perforation, arterial dissection, and embolization in a previously uninvolved vascular territory

CONTACTS AND LOCATIONS:
Overall Officials: Octavio M Pontes-Neto, MD, PhD, Principal Investigator — Hospital de Clínicas da Faculdade de Medicina de Ribeirão Preto - Universidade de São Paulo; Sheila CO Martins, MD, PhD, Principal Investigator — Hospital Moinhos de Vento; Raul G Nogueira, MD, Principal Investigator — University of Pittsburgh Medical College
Locations (13):
- Brazil (13):
  - Hospital Moinhos de Vento, Porto Alegre, Rio Grande do Sul
  - Hospital das Clínicas Botucatu, Botucatu
  - Hospital de Base do Distrito Federal, Brasília
  - Hospital das Clínicas da UFPR, Curitiba
  - Hospital Geral de Fortaleza, Fortaleza
  - Hospital de Clinicas de Porto Alegre, Porto Alegre
  - Hospital das Clínicas da Faculdade de Medicina de Ribeirão Preto, Ribeirão Preto
  - Hospital de Base de Rio Preto, São José do Rio Preto
  - Hospital das Clínicas de São Paulo, São Paulo
  - Hospital Sao Paulo, São Paulo
  - Santa Casa de Misericordia de Sao Paulo, São Paulo
  - Hospital Universitário de Uberlândia, Uberlândia
  - Hospital Estadual Central, Vitória

IPD SHARING:
Plan to Share IPD: Undecided